CLINICAL TRIAL: NCT06576791
Title: Urethral Rotation Angles and Foot Pronation Mechanical Changes in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, rovan mohamed saad elbesh, doctor, Cairo University
Other Study IDs: [P.T.REC/012/004226]
Record Dates: First submitted 2022-09-19; First posted 2024-08-29 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-06

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stress urinary incontinence (SUI) occur secondary to increased intra abdominal pressure, that directed the researchers to study the mechanical changes in urethra and bladder that associated with it. However, these urethral mechanical changes may be related to other mechanical changes in the body.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) affects about 26% of women between 30 and 59 years of age. It is the sudden involuntary urine leakage secondary to increased intra abdominal pressure related to physical activities as laughing, sneezing, straining, coughing, or exercising . There are two common mechanisms for SUI: urethral hypermobility due to loss of support of the bladder neck and urethra (affected by increased intra-abdominal pressure), and weakness of the urinary sphincter that may result from trauma, repeated urogynaecological surgeries, neurological disease, ageing or diseases leading to systemic muscular atrophy. SUI is the most common pelvic floor dysfunction linked to the vaginal delivery. However the prevalence of stress incontinence peaks occurs in the fifth decade of life . and all types of incontinence are commonly occurring with ageing and obesity.

Urethral hypermobility means that the proximal part of the urethra may exhibit a rotational movement in a postero-inferior direction. And it was diagnosed when the urethra rotated during strain over 30° from its resting axis . Urethral rotation angles may assist in both assessment and diagnosis of patients with SUI, which may in turn decreases requires for any other investigations .The ultrasonography assessment of the angle of inclination (α angle: the angle between the axis of the proximal urethra and the central axis of the symphysis pubis) and posterior urethrovesical angle (β angle: the angle between the proximal urethra and the posterior vesical wall) has been investigated by several researchers. However, recently transperineal ultrasonography is a practical, reliable, non-invasive and comfortable method for evaluation of SUI. Additionally, it has the advantage of dynamic evaluation during the Valsalva maneuver .

Urinary sphincter composed of; internal urethral sphincter that is predominantly smooth muscle without voluntary control, and the external urethral sphincter and pelvic floor muscles (PFMs) that are predominantly striated muscle with voluntary control. During activities the PFMs contract to prevent the leakage of urine, in addition, they play a significant role in trunk stabilization through its connections with abdominal muscles, diaphragm, and gluteus by myofascial continuity . Contractions of PFMs lead to activation of gluteal muscles especially the levator ani through their connection by the fossa ischioanalis . Additionally, rotators mainly the internal obturator and piriformis muscles are important for maintaining pelvic stability and PFM functionality .Moreover, the tension of the rotator cuff and gluteal muscles is also primarily determined by position of the foot. So, the tension of PFM may affect the tension and functioning of the rotators and gluteal muscles, thus influencing the biomechanics and position of whole lower limb even the foot position .

ELIGIBILITY:
Inclusion Criteria:

* multiparous vaginal delivery women
* experienced more than one delivery.

Exclusion Criteria:

* urinary tract infection
* any previous genitourinary surgery
* congenital bone deformities, pelvic organ prolapse
* taking any drugs for treating SUI
* any hormonal replacement therapy
* residual urine more than 150cc
* history of lung diseases associated with chronic coughs

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ll participants were assessed for their eligibility to participate in the study if they multiparous vaginal delivery women experienced more than one delivery with average three deliveries.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
1- Measuring urethral rotation angles by transperineally ultrasound TPUS | 3 months
  TPUS was performed using a Toshiba US machine with a 3.5 MHz electronic micro convex array probe. The bladder was comfortably partially filled with urine (about 150 mL).
2- foot pronation | 3 months
  drop test

SECONDARY OUTCOMES:
weight | 3 months
  kg

CONTACTS AND LOCATIONS:
Locations (1):
- Rovan Elbesh, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided